CLINICAL TRIAL: NCT00398983
Title: Randomized Study of Decitabine Versus Observation or Continued Standard Chemotherapy as Maintenance Therapy for Adults With Unfavorable Risk AML in First Complete Remission (CR) or Adults With Relapsed AML in Second or Greater CR
Brief Title: Randomized Study of Decitabine in Maintenance Therapy of Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0358
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Results first posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-01

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Acute Myelogenous Leukemia; AML; Remission; Decitabine; Maintenance Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decitabine 20 mg/m^2 (Experimental): 20 mg/m^2 intravenous (IV) daily for 5 days
  Interventions: Drug: Decitabine
- No Study Drug (No Intervention): Continue current therapy.

INTERVENTIONS:
Drug: Decitabine — 20 mg/m^2 IV over 1 hour daily for 5 days
  Other Names: Dacogen
  Arms: Decitabine 20 mg/m^2

SUMMARY:
The goal of this clinical study is to find out whether continued therapy with decitabine after achieving a remission in acute myeloid leukemia (AML) patients can help prolong the remission and prevent relapse of the disease.

DETAILED DESCRIPTION:
Methylation is a change that occurs to DNA that has an effect on how genes are used in human cells. It is very common in leukemias for methylation to happen abnormally. Decitabine is a new drug that blocks DNA methylation. At low doses (such as those used in this study), decitabine blocks proteins important in abnormal DNA methylation, which may, in turn, allow leukemia cells to die and disappear.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 groups. Group 1 will receive decitabine about every 4-8 weeks to see whether this drug is useful in lengthening the duration of remission in patients like you. Group 2 will not receive the study drug.

If you are assigned to Group 1, the drug will be given over about 1 hour through a peripheral or central catheter every day for 5 days. A peripheral or central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure. You will receive the study drug for 5 days per study "cycle". Each cycle will be about 4-8 weeks. You must receive your study drug at M. D. Anderson Cancer Center.

You may remain on study for up to 12 Cycles. You will be taken off study if the disease gets worse, your doctor feels it is in your best interest, or you develop intolerable side effects.

During the study, blood (about 2 tablespoons) will be drawn for routine tests every week during the first month and then every 2-4 weeks after that. You will also have a bone marrow examination aspirate/biopsy every 3-6 months to make sure that your disease remains in remission.

If you are assigned to Group 2, you will continue under the care of your doctor. This will include study visits and having a bone marrow examination aspirate/biopsy every 3-6 months up to one year after randomization to make sure that the disease remains in remission.

Once you are off study, blood (about 2 tablespoons) will be drawn and you will have a bone marrow biopsy/aspirate.

This is an investigational study. Decitabine is FDA-approved and is commercially available. It is not FDA approved for this usage, and it has been authorized for use in research only. Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years) with acute myelogenous leukemia (AML) by World Health Organization (WHO) criteria (greater than 20% blasts) and unfavorable risk cytogenetics (including intermediate and poor risk categories) in first CR or complete remission without full platelet recovery (CRp)
* Adult patients (greater than 18 years) in second or subsequent Complete Response (CR) (or CRp)
* Patients in first CR (or CRp) may have received any induction chemotherapy regimen; they may have received post-remission consolidation therapy (except for transplant) prior to inclusion in this protocol
* Patients in 2nd or subsequent CR (or CRp) may have received any appropriate salvage regimen before achieving CR and may have received further therapy before inclusion
* Performance status of 0, 1, or 2
* Adequate organ function with creatinine less than or equal to 2.0 mg/dL, bilirubin less than or equal to 3.5 mg/dL and aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) less than or equal to 3 times institutional upper limit of normal

Exclusion Criteria:

* Pregnant or lactating; women of child-bearing potential (WOCBP) must have negative pregnancy test. WOCBP defined as not post-menopausal for 12 months or no previous surgical sterilization
* Known to be HIV+
* Active and uncontrolled disease/infection as judged by the treating physician
* Unable or unwilling to sign the consent form
* No other investigational therapy within the past 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 8/28/2006 to 10/15/2009. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of the fifty participants registered, forty-five participants were evaluable. Twenty were randomized to Decitabine 20 mg/m^2, and twenty-five were randomized to no study drug. Five participants withdrew consent or developed complications before assignment of treatment.
Period: Overall Study
Arm/Group | Decitabine 20 mg/m^2 | No Study Drug
Started | 20 | 25
Completed | 20 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine 20 mg/m^2 | No Study Drug | Total
Number analyzed (Participants) | 20 | 25 | 45
Age Continuous [Median (Full Range); unit: years] | 62 [24 to 79] | 53 [31 to 72] | 57 [24 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  United States | 20 | 25 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse-Free Response at 1 Year
Description: Relapse free response defined an absence of relapse at one year of follow up.
Time Frame: Baseline to 1 year
Measure: Number; unit: participants
Arm/Group | Decitabine 20 mg/m^2 | No Study Drug
Number analyzed (Participants) | 20 | 25
participants | 10 | 10

ADVERSE EVENTS:
Time Frame: Five years, eight months.
Arm/Group | Decitabine 20 mg/m^2 | No Study Drug
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/25
Other Adverse Events (participants affected / at risk) | 20/20 | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine 20 mg/m^2 (N=20) | No Study Drug (N=25)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine 20 mg/m^2 (N=20) | No Study Drug (N=25)
Neutropenia (Blood and lymphatic system disorders) | 19 (19) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (14) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 3 (3)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No